CLINICAL TRIAL: NCT02609568
Title: Studying the Significance of Salivary Biomarkers in Pediatric Traumatic Brain Injury
Brief Title: Salivary Biomarkers in Pediatric Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Valleywise Health (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-055
Record Dates: First submitted 2014-10-16; First posted 2015-11-20 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Traumatic Brain Injury
Keywords: Children; Head injury; Salivary biomarker; Trauma Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Salivary biomarkers: S100B, neuron-specific enolase, GFAP
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control Group 1: Children with non-trauma complaints
- Control Group 2: Children with non TBI and musculoskeletal trauma
- Cases: Children admitted to hospital with moderate/severe isolatedTBI

SUMMARY:
By studying individual biomarkers in body fluids such as saliva, there is a potential for detecting injury to the brain resulting from an acute traumatic even that may not be detectable by conventional neuroimaging like CT scans.

DETAILED DESCRIPTION:
Although identification of biomarkers following TBI is a rather novel area of research, few studies that have been done in patients with severe TBI and biomarkers from serum and cerebrospinal fluid have shown to have prognostic significance. However there are no prior studies looking at biomarkers in salivary specimens. In this study we will include patients with moderate and severe TBI who require inpatient admission, and will study 3 specific salivary biomarkers. This is a unique project, since salivary specimen collection is easy and non-invasive and can be collected at any site even on a sports field by using a simple absorbable swab resembling a cigarette stub, unlike blood or CSF that can be highly invasive. Salivary specimens can also be frozen and stored for long periods of time prior to testing. If our study detects abnormalities in levels of these biomarkers when compared to healthy controls, and children with extra-cerebral injuries, in future studies we can look at children and adolescents with minor head traumas and concussions who are discharged from the emergency department after evaluation, and study their long-term outcomes and correlation with salivary biomarkers.

Specific aims:

To study levels of three specific biomarkers in salivary specimens (GFAP, S100B and NSE) in children with moderate TBI (GCS: 9-12) and severe TBI (GCS: <8) admitted to a pediatric trauma referral center. These biomarkers have been shown to have prognostic significance in prior studies using serum and CSF.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0 to 20 who present to the pediatric ED or trauma bay with an isolated acute head injury (moderate or severe) and are admitted for inpatient management;
* Pediatric patients who present to the ED with non-trauma complaints; and
* Pediatric patients who present to the ED with non-head trauma such as musculoskeletal injuries.

Exclusion Criteria:

* Patients with multisystem trauma;
* Patients with minor head trauma (GCS 13-15) discharged from the pediatric ED
* Patients with other pre-existing neurological conditions (such as cerebral palsy, chronic seizure disorder, VP shunts);
* Patients with a history suggestive of head trauma from chronic abuse;
* Incarcerated patients or patients from juvenile detention facilities;
* Refusal of parent/patient to participate for any specific reason.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1) Children aged 0 to 20 who present to the pediatric ED or trauma bay with an isolated acute head injury (moderate or severe) and are admitted for inpatient management; 2) pediatric patients who present to the ED with non-trauma complaints; and 3) pediatric patients who present to the ED with non-head trauma such as musculoskeletal injuries.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2014-04-16 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Levels of 3 specific salivary biomarkers (GFAP, S100B, and NSE) | Within 24 hours of injury
  Within 24 hours of an acute isolated TBI

SECONDARY OUTCOMES:
Glasgow Coma Scale measurement of injury severity | Day 1
  Glasgow Coma Scale is a score between 3 and 15, 3 being the worst, and 15 the best. It is composed of three parameters: Best Eye Response, Best Verbal Response, and Best Motor Response. A Coma Score of 13 or higher correlates with a mild brain injury, 9 to 12 is a moderate injury and 8 or less a severe brain injury.
Brain CT Scan abnormalities suggesting significant brain injury | Within 24 hours of injury
  Dichotomous measure: presence or absence of such abnormalities
Need for mechanical ventilation | During hospitalization (up to 50 days)
  Mechanical ventilators are used for patients who cannot breathe by themselves. Dichotomous measure: whether or not mechanical ventilation is needed.
Need for neurosurgical intervention including ICP monitor | During hospitalization (up to 50 days)
  Dichotomous measure: whether or not neurosurgical intervention is needed
Patient's Length of Stay or hospitalization | Duration of hospitalization (up to 50 days)
  Number of days spent in hospital
Final disposition | At end of hospitalization (up to 50 days)
  Polytomous measure: Discharge to home, discharge to rehab, or death

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Yeung, MD, Study Director — Valleywise Health; Kevin Foster, MD, Study Director — Valleywise Health
Locations (1):
- Maricopa Integrated Health System, Phoenix, Arizona, United States

REFERENCES:
- [Background] Zetterberg H, Smith DH, Blennow K. Biomarkers of mild traumatic brain injury in cerebrospinal fluid and blood. Nat Rev Neurol. 2013 Apr;9(4):201-10. doi: 10.1038/nrneurol.2013.9. Epub 2013 Feb 12. PMID 23399646
- [Background] Olsson B, Zetterberg H, Hampel H, Blennow K. Biomarker-based dissection of neurodegenerative diseases. Prog Neurobiol. 2011 Dec;95(4):520-34. doi: 10.1016/j.pneurobio.2011.04.006. Epub 2011 Apr 16. PMID 21524681
- [Background] Faul M, Xu L, Wald MM, Coronado V. Traumatic brain injury in the United States: emergency department visits, hospitalizations, and deaths, 2002--2006. Atlanta, GA: CDC, National Center for Injury Prevention and Control; 2010.